CLINICAL TRIAL: NCT04034264
Title: Characterization of Febrile Disease Landscape in Cambodia Via Metagenomic Pathogen Sequencing
Brief Title: Febrile Disease Landscape in Cambodia Via Metagenomic Pathogen Sequencing
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919109; 19-I-N109
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12-04

CONDITIONS: Vector-Borne Diseases; Emerging Pathogens
Keywords: Next-Generation Sequencing; Vector-Borne Diseases; Southeast Asia; Agnostic Tools; Febrile Surveillance; Natural History
MeSH Terms: conditions — Vector Borne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Afebrile close contact: Lived in the same household or worked in the same enclosed workspace daily with a febrile enrollee at the time they got sick with a known highly morbid and/or transmissible pathogen.
- Febrile patient: Patients between 2 months and 65 years old who present with fever, or diagnosed with a highly morbid and/or transmissible pathogen by clinically validated tests.

SUMMARY:
Background:

Vector-borne diseases are caused by the bite of an infected mosquito, fly, flea, tick, or other blood-feeder. These diseases cause almost 1 million deaths per year. And they are on the rise, particularly in Southeast Asia in particular. Researchers think that these diseases make up about 10 percent of fevers in Cambodia. But many of these illnesses are never diagnosed. Studying these diseases can help find new ways to identify and treat them.

Objective:

To find pathogens in people who have a fever using metagenomic pathogen sequencing platforms.

Eligibility:

People aged 2 months to 65 years with a fever of at least 38 degrees Celsius or those diagnosed with infection by a pathogen of concern who visit the referral hospital in Cambodia. Close contacts of people diagnosed with infection by a pathogen of concern may also be enrolled.

Design:

Participants will be screened with their medical history. Children will be weighed to make sure they are big enough to give blood samples.

Participants will share data about their sex, age, and where they live. They will answer more questions about their heath history. They will answer questions about and any places to which they have recently traveled. They will take a questionnaire. They will have a blood test. If they have respiratory symptoms, they will have a nasal swab.

Participants may be contacted within 1-2 weeks (early) and/or within 3 months (late) from their enrollment date to provide an optional follow-up blood samples and nasal swabs.

DETAILED DESCRIPTION:
Vector-borne diseases continue to cause significant global morbidity and mortality, particularly in Southeast Asia. However, given a lack of diagnostics available in resource-poor countries, many vector-borne diseases are never diagnosed and therefore their impact is underappreciated. Cross-sectional retrospective surveys have revealed higher than expected antibody prevalence to a number of diseases including mosquito-borne viruses and ectoparasite-borne rickettsial diseases.

Here, we aim to collect specimens from individuals with acute febrile illness or red flag pathogens to better describe the febrile disease landscape of Cambodia using novel genomics technologies (unbiased next-generation sequencing) to investigate possible infectious etiologies of illnesses of unexplained etiology in Cambodian children and adults. If a highly transmissible and/or highly virulent (red flag) pathogen of public health concern is identified, we will take a convalescent sample from the individual and screen his/her close contacts with serological and molecular assays to add an additional layer of understanding of the disease burden. With the current rise of vector-borne diseases around the world, we hope the results of this study contribute to better understanding the epidemiology and burden for

vector-borne diseases in this region.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures.
* Male or female, aged 2 months to 65 years.
* Meets one of the following case definitions:

  * Febrile patient: has documented fever equal to or greater than 38 degrees celsius in previous 24 hours.
  * Red flag patient: is an individual with disease relating to a red flag pathogen (see list, below), with confirmed standard laboratory testing (e.g., blood culture, polymerase chain reaction [PCR]) for the pathogen in question.
  * Afebrile close contact: is an afebrile individual who lived in the same household or worked in the same enclosed workspace on a daily basis with a red flag patient at the time they got sick with a known pathogen.
* Willing to allow biological samples to be stored for future research and for all de-identified metagenomic sequencing data to be stored in publicly accessible databases.

EXCLUSION CRITERIA:

* Any underlying, chronic, or current medical condition that, in the opinion of the investigator, would interfere with participation in the study (e.g., inability or great difficulty in drawing blood).
* Any febrile individual who has had surgery in the prior month.
* Any patient who enrolled and exited this study within 30 days of the initial study blood draw, or afebrile close contact who enrolled and exited within 14 days.

Ages: 2 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Febrile patients who have documented fever equal to or greater than 38 degrees celsius in previous 24 hours, or those with a highly morbid and/or transmissible pathogen detected using standard clinical tests, who present at a hospital. If there is a highly morbid and/or transmissible pathogen identified from the febrile patient, close contacts will be identified through discussion with the patient.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Identification of pathogen sequences | Enrollment (between Day 0-2)
  This is an attempt to characterize what fraction of unexplained febrile illness is vector-borne in peri-urban Cambodia. Data from this study will be used to guide future studies.

SECONDARY OUTCOMES:
Assessment of reactivity to salivary gland homogenate reactivity of appropriate vector as detected by ELISA or Western blot assays. | Enrollment (between Day 0-2)
  Characterizing vector salivary protein reactivity profiles (mosquitos, ticks, fleas) in Cambodians with vector-borne disease is the first step to better understanding transmission patterns, responsible vectors, and Cambodian people s risk of exposure to these vectors.

CONTACTS AND LOCATIONS:
Overall Officials: Christina C Yek, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (6):
- Cambodia (6):
  - Kampong Speu Referral Hospital, Chbar Mon
  - Kantha Bopha Hospital, Phnom Penh
  - Khmer-Soviet Friendship Hospital, Phnom Penh
  - National Pediatric Hospital, Phnom Penh
  - Preah Kossomak Hospital, Phnom Penh
  - Takeo District Referral Hospital, Takeo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vong S, Khieu V, Glass O, Ly S, Duong V, Huy R, Ngan C, Wichmann O, Letson GW, Margolis HS, Buchy P. Dengue incidence in urban and rural Cambodia: results from population-based active fever surveillance, 2006-2008. PLoS Negl Trop Dis. 2010 Nov 30;4(11):e903. doi: 10.1371/journal.pntd.0000903. PMID 21152061
- [Background] Gu W, Miller S, Chiu CY. Clinical Metagenomic Next-Generation Sequencing for Pathogen Detection. Annu Rev Pathol. 2019 Jan 24;14:319-338. doi: 10.1146/annurev-pathmechdis-012418-012751. Epub 2018 Oct 24. PMID 30355154
- [Background] Tabor A, Valle MR. Report from the 'One Health' 9th Tick and Tick-Borne Pathogen Conference and the 1st Asia-Pacific Rickettsia Conference, Cairns, Australia, 27th August-1st September 2017. Vet Sci. 2018 Oct 2;5(4):85. doi: 10.3390/vetsci5040085. PMID 30279400